CLINICAL TRIAL: NCT00427453
Title: A Phase I Study of the Safety and Immunogenicity of a Recombinant MVA Vaccine Encoding a Secreted Antigen From M. Tuberculosis, Antigen 85A, Delivered Intradermally by a Needle Injection in Healthy Volunteers Who Have Received BCG Immunisation 1 Month Previously
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB004
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2006-12

CONDITIONS: Tuberculosis
Keywords: Mycobacterium tuberculosis; 85A antigen; Recombinant Modified Vaccinia Virus Ankara; Phase I study; Immunogenicity; BCG
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

INTERVENTIONS:
Biological: MVA85A

SUMMARY:
This is a phase I study to test the immunogenicity of a recombinant vaccine based on Modified Vaccinia Ankara (MVA) expressing the antigen 85A (from Mycobacterium tuberculosis). This vaccine is delivered intradermally by a needle injection in healthy volunteers previously vaccinated with BCG.

DETAILED DESCRIPTION:
This is a phase I study to test the immunogenicity of a recombinant vaccine based on Modified Vaccinia Ankara (MVA) expressing the antigen 85A (from Mycobacterium tuberculosis). This vaccine is delivered intradermally by a needle injection in healthy volunteers who have recieved a BCG immunisation month previously.

1. Selection of volunteers

   Volunteers for the study will be recruited through advertisements. Each volunteer will have received an information sheet concerning the study and will have agreed to participate in writing. Volunteers will be given at least 48 hours between reading the information leaflet and agreeing to participate. Female volunteers will be told of the theoretical risk of congenital anomaly should they become pregnant during the study and only those who undertake to take precautions to avoid pregnancy during the study period will be eligible. Volunteers will give signed consent for their GP's to be notified about their participation in the trial. The GP will be faxed a letter on the day of screening and asked to reply if they know of a reason why the volunteer should not take part. The signed consent form will also be faxed with the letter.
2. Screening

   Volunteers will be asked to sign the informed consent form for screening. The following will be performed:
   * Medical history and examination
   * Laboratory evaluations - including clinical chemistry, haematology, HLA typing, anti-vaccinia antibodies, anti-HBV antibodies, anti-HCV antibodies, anti-HIV antibodies
   * Heaf test - to exclude prior exposure to TB
   * Urinalysis and urine pregnancy test if female
3. Inclusion Criteria

   * Healthy adult aged 18-55 years.
   * Normal medical history and physical examination.
   * Normal urine dipstick, blood count, liver enzymes, and creatinine.
4. Exclusion Criteria

   1. Exposure to TB/BCG vaccination at any point. Previous residence in a TB endemic area.
   2. Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
   3. Oral or systemic steroid medication or the use of immunosuppressive agents.
   4. Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
   5. Heaf test greater than Grade 0
   6. Confirmed pregnancy
   7. Previous MVA immunisations
5. Withdrawal Criteria

   1. Withdrawal of consent by subject for any reason
   2. Loss to follow-up
   3. Non-compliance with study procedures
   4. Protocol violation
   5. Serious adverse event (as defined in Appendix 3)
   6. Any other reason at discretion of the Principal Investigator
   7. Confirmed pregnancy during study period
6. Immunisation

   On Day 0, subjects will receive a single intradermal injection of 0.1ml BCG (SSI strain) over the deltoid muscle. Blood will be taken at 2 weeks and 4 weeks after this immunisation. At 4 weeks, after blood has been taken, volunteers will be immunised with 5 x 107pfu MVA85A in 0.1ml. Subjects will be observed for an hour after MVA85A immunisation. Vital signs will be monitored at 30 and 60 minutes post-immunisation. Local reactions at the site of administration will be evaluated at 60 minutes.

   A photograph of the injection site may be taken at 48 hours (with written consent). The injection site will be reviewed 7 days after each immunization.

   Blood will be taken at the following time points: At the screening visit*, prior to the BCG vaccination, 2 weeks and 4 weeks after BCG, *1 week after the MVA85A vaccination, 2 weeks, 4 weeks, *8 weeks, and *24 weeks after the vaccination. Up to 55 mls will be taken at any one time with the total being no more than 500 mls over the study period. *Samples taken on these dates will be tested for full blood count and biochemical screen. Immunological assays will be performed at all time points to determine vaccine immunogenicity. A pregnancy test will be performed prior to vaccination for female volunteers. Peripheral blood mononuclear cells will be prepared for cellular immunological assays to be performed without or following cryopreservation. Other serological measures of immune response, i.e. antibody titres, will be assayed on frozen plasma samples.

   All blood tests will be taken within 1-3 days of the due date as described in the schedule above.
7. Endpoints

The occurance and severity of local side-effects The occurance and severity of systemic side-effects The induction of T cell responses (as measured by an interferon-gamma Elispot assay).

Proliferation assays and cytotoxic T cell assays will be performed on strong CD4+ and CD8+ responses respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-55 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

Exclusion Criteria:

* Exposure to TB/BCG vaccination at any point. Previous residence in a TB endemic area.
* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Oral or systemic steroid medication or the use of immunosuppressive agents.
* Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
* Heaf test greater than Grade 0
* Confirmed pregnancy
* Previous MVA immunisations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-06; Study Completion 2005-03

PRIMARY OUTCOMES:
The occurance and severity of local and systemic side effects will be monitored. Vital signs and local reactions will be monitored at 30 and 60 minutes after each mmunisation (and after 7 days).
Blood will be taken at: the screening visit, prior to the BCG vaccination, 1 and 4 weeks after the BCG vaccination, and also at 1,4, 8, 12 and 24 weeks after the MVA85A vaccination.

SECONDARY OUTCOMES:
Immunogenicity will be measured: The induction of T cell responses (as measured by an interferon-gamma Elispot assay) will be performed on PBMCs from blood samples taken at the specified time points.
Proliferation assays and cytotoxic T cell assays will be performed. Other serological measures of immune response, i.e. antibody titres will be analysed on frozen plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, MD and PhD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Pathan AA, Sander CR, Fletcher HA, Poulton I, Alder NC, Beveridge NE, Whelan KT, Hill AV, McShane H. Boosting BCG with recombinant modified vaccinia ankara expressing antigen 85A: different boosting intervals and implications for efficacy trials. PLoS One. 2007 Oct 24;2(10):e1052. doi: 10.1371/journal.pone.0001052. PMID 17957238